CLINICAL TRIAL: NCT00231231
Title: Carotid Artery Stenting With Emboli Protection Surveillance-Post-Marketing Study (CASES-PMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04-5204
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: -PRECISE Nitinol Stent System (5F, 5.5F and 6F)
Device: ANGIOGUARD™ XP Emboli Capture Guidewire (ECGW)

SUMMARY:
The primary objective of this study is to assess the outcomes of stenting with distal protection in the treatment of obstructive carotid artery disease during peri-approval/initial commercialization in relation to the outcomes of the Sapphire Clinical Trial. The devices to be utilized are the Cordis PRECISE Nitinol Stent Systems and the Cordis ANGIOGUARD™ XP Emboli Capture Guidewire (ECGW).

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be > 18 years of age.
2. The patient has a 50% stenosis (as determined by ultrasound or angiogram) of the common or internal carotid artery and is clinically symptomatic; i.e., within the previous 180 days has experienced symptoms in the ipsilateral carotid artery distribution, defined as:

   * one or more TIAs, characterized by distinct focal neurologic dysfunction or monocular blindness with clearing of signs and symptoms within 24 hours, or
   * one or more completed strokes (as defined by this protocol) with persistence of symptoms or signs for more than 24 hours (the most recent event is used as the qualifying event), except as excluded below, with stenosis >50%, (as determined by ultrasound or angiogram) of the common or internal carotid artery, OR The patient must have a >80% diameter stenosis (as determined by ultrasound or angiogram) of the internal or common carotid artery without neurological symptoms.
3. To be entered into the study, the patient must have one or more of the following conditions:

   · congestive heart failure (class III/IV) and/or known severe left ventricular dysfunction LVEF < 30%
   * open heart surgery within six weeks
   * recent MI (>24 hours and <4 weeks)
   * unstable angina (CCS class III/IV)
   * synchronous severe cardiac and carotid disease requiring open heart surgery and carotid revascularization
   * severe pulmonary disease to include any of the following:

<!-- -->

1. chronic oxygen therapy
2. resting PO2 of 60 mmHg
3. baseline hematocrit 50%
4. FEV1 or DLCO 50% of normal. · contralateral carotid occlusion · contralateral laryngeal palsy · post-radiation treatment · previous CEA recurrent stenosis · high cervical ICA lesions · CCA lesions below the clavicle · severe tandem lesions

   * abnormal stress test.

4. The qualifying ultrasound or angiogram was performed less than 30 days prior to study entry.

· Stenosis >50%: PSV>130 cm/sec; EDV <135 cm/sec

· Stenosis >80%: PSV>220 cm/sec; EDV <135 cm/sec

· PSV ICA/PSV CCA ratio 4.0

5. The target vessel is in the native common or internal carotid artery. The arterial segment to be treated has a diameter between 4 mm and 9 mm as the largest diameter either proximal or distal to the lesion.

Exclusion Criteria:

1. The patient is experiencing an acute ischemic neurologic stroke or has experienced a stroke within the past 48 hours.
2. There is any visual angiographic or ultrasound evidence of intraluminal thrombus thought to increase the risk of plaque fragmentation and distal embolization.
3. There is total occlusion of the target carotid artery treatment site.
4. The reference segment diameter (distal common carotid and internal carotid artery segment cephalic to the lesion) is less than 4mm or greater than 9mm. See Instructions For Use, for proper stent sizing. The exception to this would be with a lesion having >95% stenosis where the true diameter of the distal vessel cannot be determined such as the case with a string sign or distal vessel collapse. In this case the judgment of the interventionalist will prevail with the intention not to oversize the stent to the distal vessel by more than 2mm.
5. The patient has any intracranial aneurysm (> 9 mm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is a 30-day composite of major adverse clinical events (MAE) including any death, myocardial infarction, or stroke. | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Sidney A. Cohen, MD, PhD, Study Director — Cordis US Corp.
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Result] Katzen BT, Criado FJ, Ramee SR, Massop DW, Hopkins LN, Donohoe D, Cohen SA, Mauri L; CASES-PMS Investigators. Carotid artery stenting with emboli protection surveillance study: thirty-day results of the CASES-PMS study. Catheter Cardiovasc Interv. 2007 Aug 1;70(2):316-23. doi: 10.1002/ccd.21222. PMID 17630678
- [Derived] Schreiber TL, Strickman N, Davis T, Kumar V, Mishkel G, Foster M, Donohoe D, Britto S, Ansel G; CASES-PMS Investigators. Carotid artery stenting with emboli protection surveillance study: outcomes at 1 year. J Am Coll Cardiol. 2010 Jun 29;56(1):49-57. doi: 10.1016/j.jacc.2010.02.045. PMID 20620717